CLINICAL TRIAL: NCT06108492
Title: A Phase I Clinical Study of SHR-2005 Intravesical Instillation in the Treatment of Intermediate and High-risk Non-muscle Invasive Bladder Cancer (NMIBC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-2005-I-101
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2023-12

CONDITIONS: Intermediate and High-risk Non-muscle Invasive Bladder Cancer

STUDY DESIGN:
Intervention Model Description: This study is an open-label, multicenter Phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics and efficacy of SHR-2005 for Intravesical perfusion in patients with intermediate and high-risk non-muscle invasive bladder cancer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-2005 (Experimental): Only one arm with SHR-2005
  Interventions: Drug: SHR-2005

INTERVENTIONS:
Drug: SHR-2005 — In dose Escalation: Four dose levels are preset. The administration cycle included 6 times of induction perfusion period and 15 times of maintenance perfusion period.
  In indication Expansion: Indications will be selected to evaluate preliminary efficacy.

SUMMARY:
This study is an open-label, multicenter Phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics and efficacy of SHR-2005 for Intravesical perfusion in patients with intermediate and high-risk non-muscle invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form;
2. ≥18 years of age, either sex;
3. Previous pathological biopsy was diagnosed as intermediate or high-risk NMIBC ;
4. ECOG performance status of 0-1;
5. Life expectancy ≥ 2 years;
6. Adequate bone marrow and organ function.

Exclusion Criteria:

1. Received TURBT or other surgical treatment or radiotherapy for bladder lesions within 2 weeks before the first administration;
2. Patients who were receiving treatment in other clinical trials or less than 4 weeks from the end of the first administration in this study;
3. History of serious cardiovascular and cerebrovascular diseases;
4. Severe infection within 2 weeks prior to the first dose;
5. Adverse reactions of previous anti-tumor treatment have not recovered to Grade ≤ 1 per NCI-CTCAE v5.0;
6. Oversize surgery or severe trauma within 4 weeks before the first use of research drugs;
7. Previously received any TNFR agonist antibody therapy, such as OX40, CD137, CD27, CD357 antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | From Day 1 to Day 21
Maximum tolerated dose (MTD) | From Day 1 to Day 21
Incidence and severity of adverse events (AEs) ([CTCAE] v5.0) | From Day 1 to 90 days after last dose
RP2D（Recommended Phase 2 dose） | From Day 1 to 90 days after last dose

SECONDARY OUTCOMES:
PK parameter: Tmax of SHR-2005 | approximately 24 months
  Time to maximum concentration of SHR-2005
PK parameter: Cmax of SHR-2005 | approximately 24 months
  Maximum concentration of SHR-2005
PK parameter: AUC0-∞ of SHR-2005 | approximately 24 months
  area under the concentration-time curve from time 0 to infinity of SHR-2005
Immunogenicity of SHR-2005 | approximately 24 months
  Anti- SHR-2005 antibody (ADA)
Duration of response (DoR) | approximately within 36 months
  Evaluated using RECIST 1.1
Disease control rate (DCR) | approximately within 36 months
  Evaluated using RECIST 1.1
Progression-free survival (PFS) | approximately within 36 months
  Evaluated using RECIST 1.1
Amount_recovered and Percent_recovered | approximately 24 months
  The Amount _ recovered and Percent _ recovered of SHR-2005 in urine after intravesical instillation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided